CLINICAL TRIAL: NCT04664361
Title: Randomized, Double-blind, Placebo-controlled Clinical Trial of Nicotinamide Mononucleotide on Muscle Recovery and Physical Capacity in Healthy Volunteers With Moderate Physical Activity
Brief Title: Effect of NMN on Muscle Recovery and Physical Capacity in Healthy Volunteers With Moderate Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seneque SA (Industry)
Collaborators: CEN Nutriment (Unknown); Centre d'Expertise de la Performance (Unknown); LGD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: C1598
Record Dates: First submitted 2020-12-10; First posted 2020-12-11 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Physical Activity; Muscle Recovery
Keywords: Nicotinamide mononucleotide; Muscle pain
MeSH Terms: conditions — Motor Activity; Myalgia | interventions — Nicotinamide Mononucleotide

STUDY DESIGN:
Intervention Model Description: Randomized double-blind, placebo-controlled clinical trial conducted on 3 parallel groups
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NMN 250 (Experimental): NMN tablet (250 mg)
  Interventions: Dietary Supplement: Nicotinamide mononucleotide
- NMN 500 (Experimental): NMN tablet (500 mg)
  Interventions: Dietary Supplement: Nicotinamide mononucleotide
- Placebo (Placebo Comparator): NMN-free placebo tablet.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Nicotinamide mononucleotide — Daily supplementation with NMN at 250 and 500 mg for 38 days in total
  Arms: NMN 250; NMN 500
Other: Placebo — Daily supplementation with placebo for 38 days in total
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of NMN supplementation (250 and 500 mg/day over 38 days) compared to placebo in healthy volunteers with moderate physical activity on muscle recovery, physical capacity, cardiorespiratory recovery, the perception of the arduousness of the effort, the variation in blood lactate levels before and after physical exercise, the perception of the intensity of post-exercise muscle pain (cramps), the body composition and Nicotinamide-Adenine Mononucleotide (NAD+) level in blood.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index ranging from 20 to 28 kg/m2(bounds included);
* Body weight between of 70 kg to 100 kg (including limits);
* Able to provide written informed consent to participate;
* Having a moderate level of physical activity according to the Global Physical Activity Questionnaire (GPAQ);
* Having a sport practice involving endurance or split races (including collective or individual sports) or cycling.
* Agreeing not to change their physical activity habits throughout the study;

Exclusion Criteria:

* Having a mental state that does not allow them to give free and informed consent to participate in the study;
* Being taking regularly or have taken within the last month any medication or dietary supplement that may increase endurance, recovery, or physical capacity. In particular, the following drugs are strictly prohibited: beta-2 agonists such as salbutamol (Ventolin®), terbutaline (Bricanyl®), fenoterol (Berotec®), salmeterol (Serevent®) and formoterol (Foradil®) as well as corticosteroids;
* Having history of a recent (less than 3 months) lower extremity muscle injury;
* Presenting a depressive syndrome;
* Presenting, in the opinion of the investigator, any symptomatology, pathology or cardiovascular risk factors that are incompatible with the conduct of the study or with the performance of a stress test or that could influence the results of the study, and in particular: 1) an abnormal resting and/or stress ECG at the inclusion visit according to the investigator; 2) presence of abnormalities in the lipid balance (Total Cholesterol, Triglycerides, HDL, LDL), blood glucose, and/or hemodynamic parameters;
* Presenting an abnormal biological balance (Creatinine, Uric acid, Troponin, Alanine aminotransferase / Aspartate aminotransferase, Lactate dehydrogenase, Creatine Kinase, C-reactive protein, Transferrin, Bilirubin, Gamma Glutamyl transpeptidase, Cholesterol (EAL), Glycemia, Ionogram, Alkaline phosphatase );
* Being not be compliant with the constraints imposed by the protocol;
* Having an allergy or a contraindication to the components of the studied products;
* Being already involved in another clinical trial or being in the exclusion period of a previous clinical trial;
* Being unable to understand, speak and read French fluently;
* Being not affiliated with a health insurance company;
* Being vulnerable persons or persons deprived of liberty by a judicial or administrative decision;
* Consuming illegal psychotropic substances or having an alcohol consumption of more than 2 glasses of alcohol/wine per day.

Ages: 20 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 131 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Evolution of muscle recovery | before and after 21 and 38 days of treatment
  Wingate Anaerobic Test (WANT) preformed post-endurance test (at 85% maximum aerobic speed)

SECONDARY OUTCOMES:
Changes in physical capacity | before and after 21 and 38 days of treatment
  physical capacity evaluated during an endurance test (at 85% maximum aerobic speed) by the maximum duration (time limit)
Changes in cardiorespiratory recovery | before and after 21 and 38 days of treatment
  Measurement of blood pressure and heart rate at rest and at intervals of several minutes after the endurance test (at 85% maximum aerobic speed)
Changes in the perception of the arduousness of the effort | before and after 21 and 38 days of treatment
  evaluated by the Borg scale during the endurance test (at 85% maximum aerobic speed)
Changes in blood lactate levels before and after physical exercise | before and after 21 and 38 days of treatment
  blood lactate levels before and after the endurance test (at 85% maximum aerobic speed)
Changes in the perception of the intensity of post-exercise muscle pain (cramps) | before and after 21 and 38 days of treatment
  post-exercise muscular pain in evaluated using a 7 points numerical scale, 24, 48 and 72 hours after the endurance test
Changes in the body composition | before and after 21 and 38 days of treatment
  fat mass, muscle mass, visceral fat, water mass determined by Bioelectrical Impedance Analysis (BIA)
Changes blood NAD+ levels | before and after 21 and 38 days of treatment
  Evaluation of cellular NAD+ concentration in blood from baseline to the end of study

CONTACTS AND LOCATIONS:
Overall Officials: Nadège PLAZA, MD, Principal Investigator — CEN Nutriment
Locations (1):
- CEN Nutriment, Dijon, France

IPD SHARING:
Plan to Share IPD: Undecided